CLINICAL TRIAL: NCT01145118
Title: Reliability of Functional Outcome Measures in Plantar Fascitis Patients
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL., Clalit Health Services
Other Study IDs: K-10-0037-ctil
Record Dates: First submitted 2010-05-24; First posted 2010-06-16 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; Physiotherapy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Plantar Fasciitis (PF) is the most common foot condition treated by healthcare providers, striking approximately 2 million Americans each year. Nevertheless its causes are still not known. The risk factors for PF are known and the diagnosis, which is based on clinical assessment, is relatively simple. Still most of the treatments for PF focus on short term symptoms relief instead of prevention or reduction of recurrence.

Physical therapy treatment that focuses on reducing the symptoms for the long run and prevention, should include outcome measures, which if found to be reliable, will make the diagnosis clearer. Diagnosis based on reliable clinical and functional measures will assist the physical therapist to understand the major deficiencies of the patient, and accordingly to help him to make the right decision in choosing treatment. Also comprehensive knowledge of the characteristics of PF may enable selection of appropriate preventive measures.

DETAILED DESCRIPTION:
Objectives:

Characterize the unilateral PF syndrome using functional outcome measures, while comparing them to the healthy foot of the same patient. In addition the study will investigate the reliability of these functional outcome measures in PF patients.

Methodology:

Individuals referred to physiotherapy for PF will be assessed for eligibility and consent for the study. They will undergo two evaluations on the same week to evaluate the test- retest reliability of the functional measurements.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral plantar fasciitis
* Painful first step in the morning
* Calcaneal soreness in palpation
* Insured by Clalit Health Care Services
* Signed informed consent

Exclusion Criteria:

* Ankle or foot surgery
* Congenital deformation of foot
* Lower limb spasticity
* Using assistive devices
* Bilateral plantar fasciitis
* Refuse to participate or sign informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred to community physiotherapy center for plantar Fasceitis treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Functional Limitation | 1 week
  Measurement of Functional Limitation using Foot Function Index (FFI) compared to the healthy foot

SECONDARY OUTCOMES:
Pain intensity | 1 week
  Measurement of pain intensity using visual analog scale (VAS), compared to the healthy foot
Pain threshold | 1 week
  Measurement of pain threshold using a Pressure Algometer, compared to the healthy foot
Muscle strength | 1 week
  Measurement of Muscle strength in Plantar Flexion and Dorsi Flexion using Hand Held Dinamometer - compared to the healthy foot.
Range of motion | 1 week
  Measurement of Range of motion using a Digital inclinometer - compared to the healthy foot

CONTACTS AND LOCATIONS:
Overall Officials: Uzi Milman, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; HASAN KHAIRELDIN, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; SHARON ISRAELY, BA, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel